CLINICAL TRIAL: NCT05866003
Title: tDCS During Contralaterally Controlled FES for Upper Extremity Hemiplegia
Brief Title: tDCS + CCFES-mediated Functional Task Practice for Post-stroke Upper Extremity Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, David Cunningham, Assistant Professor, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000229
Record Dates: First submitted 2023-04-14; First posted 2023-05-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Upper Extremity Paresis; Hemiplegia
Keywords: Stroke; Rehabilitation; Therapy; Electrical Stimulation; Brain stimulation; Hand; CCFES; Motor Cortex; TMS; Motor Recovery; Central Nervous System; CVA; Upper Limb
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active conventional tDCS plus CCFES (Active Comparator): The conventional tDCS montages involves placing the surface anode electrode on the scalp of the lesioned hemisphere and the surface cathode electrode on the scalp of the non-lesioned hemisphere. TDCS will deliver a low current while participants are undergoing CCFES-mediated functional task practice.
  Interventions: Device: Active conventional tDCS montage plus CCFES; Behavioral: CCFES with Occupational Therapy
- Active unconventional tDCS plus CCFES (Active Comparator): The unconventional tDCS montages involves placing the surface anode electrode on the scalp of the non-lesioned hemisphere and the surface cathode electrode on the scalp of the lesioned hemisphere. TDCS will deliver a low current while participants are undergoing CCFES-mediated functional task practice.
  Interventions: Device: Active unconventional tDCS montage plus CCFES; Behavioral: CCFES with Occupational Therapy
- Sham tDCS plus CCFES (Sham Comparator): The sham tDCS montages involves placing the surface electrodes on the scalp over the lesioned and the non-lesioned hemisphere. TDCS will not be delivered during CCFES-mediated functional task practice.
  Interventions: Device: Sham tDCS plus CCFES; Behavioral: CCFES with Occupational Therapy

INTERVENTIONS:
Device: Active conventional tDCS montage plus CCFES — tDCS is a non-invasive brain stimulation technique. A small machine (9-volt battery operated device) will use a weak amount of electric current to stimulate the brain without any invasive procedure. Electrodes, covered in sponges soaked in saline, will be placed over certain parts of your head and held in place using a rubber strap. In addition, an electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract.
  Arms: Active conventional tDCS plus CCFES
Device: Active unconventional tDCS montage plus CCFES — tDCS is a non-invasive brain stimulation technique. A small machine (9-volt battery operated device) will use a weak amount of electric current to stimulate the brain without any invasive procedure. Electrodes, covered in sponges soaked in saline, will be placed over certain parts of your head and held in place using a rubber strap. In addition, An electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract.
  Arms: Active unconventional tDCS plus CCFES
Device: Sham tDCS plus CCFES — An electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract. The stimulator can be programmed to deliver stimulation with an intensity that corresponds to the opening of a glove instrumented with sensors and plugged into the stimulator.
  Arms: Sham tDCS plus CCFES
Behavioral: CCFES with Occupational Therapy — An electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract. The stimulator can be programmed to deliver stimulation with an intensity that corresponds to the opening of a glove instrumented with sensors and plugged into the stimulator. During the lab visits, all participants will use CCFES to assist hand opening during occupational therapy task practice.

SUMMARY:
After a stroke, it is very common to lose the ability to open the affected hand. Occupational and physical rehabilitation therapy (OT and PT) combined with non-invasive brain stimulation may help a person recover hand movement.

The purpose of this study is to compare 3 non-invasive brain stimulation protocols combined with therapy to see if they result in different amounts of recovery of hand movement after a stroke.

DETAILED DESCRIPTION:
This study is a randomized clinical trail (RCT) of stroke survivors with chronic (6 to 24 months) hemiplegia randomized to: 1) conventional transcranial direct current stimulation (tDCS), 2) unconventional tDCS, or 3) sham tDCS during contralaterally controlled functional electrical stimulation mediated occupational therapy. The treatment will last 12 weeks and be followed by a 6-month follow-up period. Assessors, therapists and participants will be blinded to which tDCS treatment is received. This will be the first RCT of tDCS + CCFES.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 and ≤ 90
2. ≥ 6 and ≤ 24 months since first clinical hemorrhagic or nonhemorrhagic stroke
3. Able to follow 3-stage command
4. Able to remember 2 of 3 items after 30 minutes
5. Full volitional elbow extension/flexion and hand opening/closing of unaffected limb
6. Adequate active movement of shoulder and elbow to position the paretic hand in the workspace for table-top task practice
7. Patient must be able to sit unassisted in an armless straight-back chair for the duration of the screening portion of the eligibility assessment
8. Medically stable
9. ≥ 10° finger and wrist extension
10. Skin intact on hemiparetic arm, hand and scalp
11. Muscle contraction can be elicited with Transcranial Magnetic Stimulation
12. Unilateral upper limb hemiparesis with finger extensor strength of ≤ grade 4/5 on the Medical Research Council (MRC) scale
13. Score of ≥1/14 and ≤ 11/14 on the hand section of the upper extremity Fugl-Meyer Assessment
14. While relaxed, surface NMES of finger extensors and thumb extensors and/or abductors produces a functional degree of hand opening without pain.

Exclusion Criteria:

1. Co-existing neurological condition other than prior stroke involving the hemiparetic upper limb (e.g., peripheral nerve injury, PD, SCI, TBI, MS).
2. Uncontrolled seizure disorder
3. Use of seizure lowering threshold medications and the discretion of the study physician
4. Cardiac pacemaker or other implanted electronic device
5. Pregnant
6. IM Botox injections in any UE muscle in the last 3 months
7. Insensate arm, forearm, or hand
8. Deficits in communication that interfere with reasonable study participation
9. Severely impaired cognition and communication
10. Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
11. Severe shoulder or hand pain (unable to position hand in the workspace without pain)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Box and Blocks Test (BBT) | Change in BBT will be assessed at 6 weeks, 12 weeks, 24 weeks, and 36 weeks
  The BBT counts how many blocks a patient can pick up, move over a barrier, and release in 60 seconds.

SECONDARY OUTCOMES:
Upper Extremity Fugl-Meyer Assessment (UEFM). | Change in UEFM will be assessed at 6 weeks, 12 weeks, 24 weeks, and 36 weeks
  The UEFM is a reliable and valid measure of post-stroke upper limb motor impairment

OTHER OUTCOMES:
Neurophysiologic Assessments | Change in neurophysiologic assessments will be assessed at 6 weeks, 12 weeks, 24 weeks, and 36 weeks
  Neurophysiologic assessments will be performed using TMS. Measures of excitability and inhibition will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: David A Cunningham, PhD, Principal Investigator — MetroHealth Medical Center and Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No